CLINICAL TRIAL: NCT00006058
Title: Study of the Pathobiology of Bronchopulmonary Dysplasia in Newborns
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital of Philadelphia (Other)
Other Study IDs: NCRR-M01RR00240-1630; CHP-IRB-97-1200; CHP-GCRC-1630
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; cardiovascular and respiratory diseases; neonatal disorders; rare disease; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Create a clinical sample bank of neonates with lung disease to test hypotheses regarding the pathogenesis of bronchopulmonary dysplasia (BPD).

II. Determine whether a developmental deficiency of surfactant protein B (SP-B) contributes to the occurrence of respiratory distress and BPD in these patients.

III. Study metabolic abnormalities associated with inherited deficiency of SP-B in these patients.

IV. Determine whether plasma nitrotyrosine levels, a marker of peroxynitrite mediated oxidant stress, are elevated in premature infants who develop BPD.

V. Measure the temporal changes in critical components of the inflammatory process (cell composition, inducible nitric oxide synthase, hyaluronan (HA), receptor for HA mediated mobility, and selected cytokines) in bronchoalveolar lavage, blood, and urine samples obtained from these patients, and to correlate these changes with their clinical course.

VI. Examine changes in the insulin-like growth factor axis that occur in the lungs of infants with respiratory distress syndrome (RDS) and BPD.

VII. Determine the relationship between degradation of elastin and the clinical course of BPD.

VIII. Determine whether the normal fall in plasma endothelin-1 concentrations after birth are delayed in infants with RDS and BPD.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Bronchoalveolar lavage and urine samples are obtained from patients on day of life 0, 1, 3, 7, 14, 21, and 28, and every 2 weeks thereafter until the infant is extubated. Serial blood samples are obtained from patients on day of life 0 (cord blood if possible), 1, 3, 7, 14, and 28, and prior to hospital discharge. Infants who require supplemental oxygen beyond 28 days of life will have 3 additional blood samples obtained at 6, 8, and 12 weeks of life. Those infants with established bronchopulmonary dysplasia who are admitted to the hospital at over 4 weeks of age have plasma samples obtained at the time of admission, and every 2 weeks thereafter for a maximum total of 5 samples.

ELIGIBILITY:
Premature infants with gestational age of less than 33 weeks requiring mechanical ventilation

OR

Term or near term infants, at least 33 weeks gestation, with severe respiratory distress, requiring mechanical ventilation with an FiO2 greater than 0.5 and mean airway pressure greater than 10

OR

Infants over 4 weeks old with established bronchopulmonary dysplasia requiring mechanical ventilation

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1996-09

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A. Ballard, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States